CLINICAL TRIAL: NCT00781248
Title: Evaluation of Safety and Efficacy of the NasoGastric Shield (NG Shield) in Healthy Subjects With Indwelling Nasogastric Tube
Brief Title: Safety and Efficacy Study of the NG Shield, a Device Intended to Reduce Pain and Discomfort Level Related to Nasogasstric Tube Usage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nanovibronix (Industry)
Responsible Party: Dr. Dagan Harris VP Clinical Affairs, NanoVibronix
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: NV-NGS-06-001
Record Dates: First submitted 2008-10-26; First posted 2008-10-28 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Intubation, Nasogastric
Keywords: enteral feeding; Subject who requires nasogastric tube

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): starting with active NG Shield
  Interventions: Device: NG Shield
- 2 (Experimental): Starting with inactive NG Shield
  Interventions: Device: NG Shield

INTERVENTIONS:
Device: NG Shield — A device to reduce pain/discomfort related to nasogastric tube usage

SUMMARY:
The purpose of the study i to demonstrate the safety and efficacy of a device that intends to reduce pain/discomfort related to nasogfastric tube usage by reducing the friction between the tube and internal orifice (nose and pharynx)using micro vibrations

ELIGIBILITY:
Inclusion Criteria:

1. Subject is in good health and able to undergoes the NG tube insertion procedure, according to the PI decision
2. Subject is able to understand and answer the pain and discomfort questionnaires
3. Subject has been fasting for at least 12h prior to the insertion phase
4. Subject underwent a physical examination by the PI
5. Subject able, agrees and signs the Inform Consent Form (ICF)

Exclusion Criteria:

1. Subject has any history of dysphagia or esophageal disease
2. Subject used anti pain medications during the last week prior to the study date
3. Subject used Antibiotics during the last week prior to the study date
4. Subject with Asthma
5. Subject with chronic or acute nasal or throat disorder
6. Subject who suffered from upper respiratory infection at least 7 days prior to the insertion procedure
7. Any pain from other source prior to the initiation of the study procedure according to the PI judgment and decision
8. Subject has any condition, which precludes compliance with study and/or device instruction for use
9. Subject is currently participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain/discomfort levelusing flicker scale (1-10 scale)during indwelling phase | every 30 minutes for 6 hours
safety of device usage | 6 hours

SECONDARY OUTCOMES:
pain/Dicomfort during insertion and removal of the nasogastric tube | at t=0h and t=6h

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Adler, M.D, Principal Investigator — "Bikur Cholim" Hospital, Jerusalem ISRAEL
Locations (1):
- "Bikur Cholim" Hospital, Jerusalem, Israel